CLINICAL TRIAL: NCT00125983
Title: A Phase II Pharmacokinetic Study of the Transdermal Contraceptive System and Oral Contraceptive in HIV-1 Infected Women on Lopinavir/Ritonavir
Brief Title: Drug Interactions Between Lopinavir/Ritonavir and Oral or Patch Contraceptives in HIV Infected Women
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: National Institute of Allergy and Infectious Diseases (NIAID) (NIH)
Collaborators: Advancing Clinical Therapeutics Globally for HIV/AIDS and Other Infections (Network)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Prevention
Other Study IDs: A5188; 10011 (Registry Identifier: DAIDS ES); AACTG A5188
Record Dates: First submitted 2005-07-29; First posted 2005-08-02 (Estimated); Last update posted 2021-11-01 (Actual); Status verified 2021-10

CONDITIONS: HIV Infections; Pregnancy
Keywords: Birth Control Pills; Oral Contraceptives; Contraceptive Patch; Pharmacokinetics; Antiretroviral Therapy, Highly Active; Protease Inhibitor; Treatment Experienced; Treatment Naive; Contraception
MeSH Terms: conditions — HIV Infections | interventions — Lopinavir; ovcon 35; Ortho Evra

INTERVENTIONS:
Drug: Lopinavir/ritonavir
Drug: Ortho Novum 1/35
Drug: Ortho Evra

SUMMARY:
The purpose of this study is to examine the drug interactions between a protease inhibitor (PI)-based regimen including lopinavir/ritonavir (LPV/r) and two forms of contraceptive medications in HIV infected women.

DETAILED DESCRIPTION:
Both PIs and oral contraceptives are metabolized by the same pathway, which significantly decreases the effectiveness of oral contraceptives and limits the contraceptive choices available to HIV infected women. More effective hormonal contraceptive methods are necessary for preventing unintended pregnancy in women taking highly active antiretroviral therapy (HAART). Ortho Evra is a contraceptive patch that was approved by the FDA in 2001; it uses a transdermal contraceptive system, and higher rates of compliance have been associated with its use, compared to oral contraceptives. Because Ortho Evra is administered as a contraceptive patch worn on the skin, it may bypass the metabolic pathway common to both PIs and oral contraceptives, making it a viable contraceptive option for HIV infected women on PI-based regimens. The purpose of the study is to examine the interaction between a PI-based regimen containing LPV/r and two forms of contraceptive medications, Ortho Evra and an oral contraceptive, Ortho Novum (ON 1/35), in HIV infected women.

Participants will be enrolled in this study for 6 weeks and will be assigned to one of two study arms, depending on their HAART regimen at study entry. Participants in both arms will also be stratified by age. Arm A participants will receive 400 mg/100 mg LPV/r twice daily along with two or more nucleoside reverse transcriptase inhibitors (NRTIs). Arm B participants will receive a regimen containing only NRTIs or no HAART. HAART will not be provided by this study. All patients will receive a single dose of ON 1/35 on Day 1 and will start the Ortho Evra contraceptive patch on Day 3. A physical exam, pap smear, pregnancy test, viral load test, CD4 and CD8 counts, and blood collection will occur at or before study entry and on Day 24. Pharmacokinetic analyses will occur on Days 1 through 3, 17 through 19, and 24.

ELIGIBILITY:
Inclusion Criteria for All Participants:

* HIV infected
* CD4 count of 200 cells/mm3 or more within 45 days of study entry
* HIV-1 RNA viral load less than 55,000 copies/ml within 45 days of study entry
* Parent or guardian willing to provide informed consent
* Negative pregnancy test within 45 days of study entry
* Willing to use acceptable forms of contraception
* Agrees not to change current smoking or non-smoking habits
* Agrees not to consume caffeine on Day 1, Days 17 through 19, and Day 24 until after the last blood sample of that day is drawn
* Agrees not to consume alcohol within 48 hours of PK sampling periods
* Patients on methadone maintenance therapy should be on a stable methadone dose for at least 60 days prior to study entry and continue maintenance therapy throughout the study

Inclusion Criteria for Arm A Participants:

* Have taken LPV/r for at least 60 consecutive days prior to study entry and taken the same dose twice daily for at least 14 days prior to study entry. Women switching from capsule formulation LPV/r to new tablet formulation of 200mg/50 mg LPV/r must be taking twice-daily doses of this formulation, for a total daily dose of 800 mg/200 mg LPV/r, for at least 7 days prior to study entry.

Inclusion Criteria for Arm B Participants:

* Have not taken or currently not taking a PI- or non-nucleoside reverse transcriptase inhibitors (NNRTI-) based regimen for at least 30 days prior to study entry, and not planning on starting PIs or NNRTIs during the 6-week study period. Women who have not been on HAART for at least 30 days prior to study entry are also eligible.
* For patients not receiving HAART, documentation that they have been counseled about the benefits of HIV treatment within 90 days of study entry and have elected not to initiate therapy

Exclusion Criteria for All Participants:

* Use of systemic hormonal therapies containing estrogens, progestins, or anabolic steroids (e.g., estrogen, progesterone, oral contraceptives, Mirena [levonorgestrol] intrauterine device [IUD], Progestasert [progesterone] IUD) within 60 days of study entry
* Anabolic therapies (nandrolone decanoate or megestrol) within 60 days of study entry
* Systemic glucocorticoids within 14 days of study entry
* Certain medical conditions. More information on this criterion can be found in the protocol.
* Need for prolonged bedrest after major surgery
* Smokers of ages 35 or older
* NNRTIs within 30 days of study entry
* Nausea, vomiting, or abdominal pain of Grade 3 or higher within 30 days of study entry
* Known allergy or sensitivity to ethinyl estradiol (EE), norelgestromin (NGMN), or components of the Ortho Evra contraceptive patch
* Known allergy or sensitivity to norethindrone or components of the ON 1/35 oral contraceptive pill
* Serious illness requiring systemic treatment or hospitalization within 14 days of study entry
* Undiagnosed abnormal vaginal bleeding
* Depo-Provera (medroxyprogesterone acetate) within 180 days of study entry
* Lunelle (estradiol cypionate and medroxyprogesterone acetate) within 90 days of study entry
* Use of certain medications within 30 days of study entry
* Current drug or alcohol use or dependence that, in the opinion of the investigator, may interfere with the study
* Unable to adhere to HAART, the Ortho Evra contraceptive patch, or single dose ON 1/35 regimens

Min Age: 13 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 32 (Actual)
Dates: Study Completion 2007-01 (Actual)

PRIMARY OUTCOMES:
Days 17, 18, 19, and 24 Ortho Evra transdermal contraceptive ethinyl estradiol (EE) area under the concentration-time curve (AUC)

SECONDARY OUTCOMES:
Intensive EE AUC pharmacokinetics (PK) after single dose Ortho Novum (ON) 1/35 and after Ortho Evra administration on Days 17, 18, 19, and 24
Day 1 intensive EE AUC PK after single dose ON 1/35
Days 17, 18, 19, and 24 norelgestromin (NGMN) AUC
changes in HIV RNA viral load, CD4 and CD8 counts and their respective percentages, sex hormone binding globulin levels, and liver enzymes from baseline to Days 17, 18, 19, and 24
occurrence of nausea and vomiting, breast tenderness, headache, skin irritation, vaginal bleeding, change in weight, change in blood pressure, change in appetite, mood changes, vaginal infection, and gallbladder disease
PK parameters of LPV in Arm A at baseline and on Days 17, 18, 19, and 24

CONTACTS AND LOCATIONS:
Overall Officials: Lori Kamemoto, MD, MPH, Study Chair — Hawaii AIDS Clinical Research Program, University of Hawaii School of Medicine
Locations (9):
- United States (8):
  - USC CRS, Los Angeles, California
  - Usc La Nichd Crs, Los Angeles, California
  - University of Colorado Hospital CRS, Aurora, Colorado
  - Univ. of Hawaii at Manoa, Leahi Hosp., Honolulu, Hawaii
  - Indiana Univ. School of Medicine, Infectious Disease Research Clinic, Indianapolis, Indiana
  - Beth Israel Med. Ctr., ACTU, New York, New York
  - Weill Med. College of Cornell Univ., The Cornell CTU, New York, New York
  - Pitt CRS, Pittsburgh, Pennsylvania
- San Juan City Hosp. PR NICHD CRS, San Juan, Puerto Rico

REFERENCES:
- [Background] Mildvan D, Yarrish R, Marshak A, Hutman HW, McDonough M, Lamson M, Robinson P. Pharmacokinetic interaction between nevirapine and ethinyl estradiol/norethindrone when administered concurrently to HIV-infected women. J Acquir Immune Defic Syndr. 2002 Apr 15;29(5):471-7. doi: 10.1097/00126334-200204150-00007. PMID 11981363
- [Background] Ouellet D, Hsu A, Qian J, Locke CS, Eason CJ, Cavanaugh JH, Leonard JM, Granneman GR. Effect of ritonavir on the pharmacokinetics of ethinyl oestradiol in healthy female volunteers. Br J Clin Pharmacol. 1998 Aug;46(2):111-6. doi: 10.1046/j.1365-2125.1998.00749.x. PMID 9723818
- [Background] Audet MC, Moreau M, Koltun WD, Waldbaum AS, Shangold G, Fisher AC, Creasy GW; ORTHO EVRA/EVRA 004 Study Group. Evaluation of contraceptive efficacy and cycle control of a transdermal contraceptive patch vs an oral contraceptive: a randomized controlled trial. JAMA. 2001 May 9;285(18):2347-54. doi: 10.1001/jama.285.18.2347. PMID 11343482
- [Result] Vogler MA, Patterson K, Kamemoto L, Park JG, Watts H, Aweeka F, Klingman KL, Cohn SE. Contraceptive efficacy of oral and transdermal hormones when co-administered with protease inhibitors in HIV-1-infected women: pharmacokinetic results of ACTG trial A5188. J Acquir Immune Defic Syndr. 2010 Dec;55(4):473-82. doi: 10.1097/QAI.0b013e3181eb5ff5. PMID 20842042